CLINICAL TRIAL: NCT02632240
Title: Collagen Matrix With Tunnel Technique Compared to CTG for the Treatment of Periodontal Recessions - Randomized Clinical Trial
Brief Title: Collagen Matrix With Tunnel Technique Compared to CTG for the Treatment of Periodontal Recessions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Silesia (Other)
Responsible Party: Principal Investigator, Lukasz Gilowski, PhD DDS, Medical University of Silesia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KNW-1-072/N/3/0
Record Dates: First submitted 2015-12-13; First posted 2015-12-16 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Gingival Recession
Keywords: gingival recession; mucogingival surgery; collagen matrix; connective tissue graft; tunnel technique
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Active Comparator): Surgery:The tunnel technique for covering gingival recession. Graft: connective tissue.
  Interventions: Other: Surgery:The tunnel technique for covering gingival recession
- Study group (Active Comparator): Surgery:The tunnel technique for covering gingival recession.Graft: xenogenic collagen matrix (Mucoderm).
  Interventions: Other: Surgery:The tunnel technique for covering gingival recession

INTERVENTIONS:
Other: Surgery:The tunnel technique for covering gingival recession — The surgery starts with the sulcular incisions in the region of recessions, which enable access for the supraperiosteal preparation. The procedure is extended into the mucosal tissue using the tunneling knives. The partial-thickness flap is performed at the buccal site. Only the papillary regions are fully detached with the periosteum. The graft is placed into the tunnel and stabilized with absorbable sutures.The mobilized mucous flap is advanced coronally and stabilized with non-absorbable suspensory sutures.

SUMMARY:
The aim of this study is to compare the efficacy of dental root coverage using the tunnel technique with connective tissue graft (CTG) and the same technique with collagen matrix for treatment of multiple gingival recessions Miller Class I and II.

This study is a randomized-controlled clinical trial of 6 months duration.

DETAILED DESCRIPTION:
According to the medical databases, there are limited randomized clinical trials comparing xenogenic collagen matrix and CTG used with the tunnel technique. The collagen matrix is a possible alternative to connective tissue graft.

The purpose of this clinical study is to compare short-term (3-6 months) outcomes of a root coverage using the tunnel technique with the collagen matrix and the same technique with CTG for the treatment of multiple recessions Miller class I and II.

Twenty eight patients are enrolled in the study. Patients in the test group are treated with xenogenic collagen matrix using the tunnel technique whereas patients in the control group with CTG. Clinical recordings are obtained at baseline and after 3 and 6 months. The percentage of average recession coverage (ARC) is evaluated after 3 and 6 months after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Presence of minimum two adjacent periodontal recessions Miller class I or II and at least 2 mm recessions depth.

Exclusion Criteria:

* Approximal Plaque Index (API) > 15%,
* Sulcus Bleeding Index (SBI) > 10%,
* Systemic diseases with compromised healing potential or infectious diseases,
* Untreated periodontal conditions,
* Pregnant and lactating females.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2014-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Clinical attachment level (CAL) | 6 months
  Distance from the cemento enamel junction to the deepest point of the gingival sulcus

SECONDARY OUTCOMES:
Recession depth (RD) | 6 months
  Distance from the mid-facial point of the cemento-enamel junction to the free gingival margin
Recession width (RW) | 6 months
  Recession width horizontally at cemento-enamel junction level
Width of keratinized tissue (KTW) | 6 months
  Distance from the mucogingival junction to the gingival margin
Recession area (RA) | 6 months
  The area of a triangle with a width of recession as the base and a depth of the recession as the height.
the average percentage of root coverage (ARC) | 6 months
  The percentage of covered recession area.
The complete coverage of recessions (CRC) | 6 months
  The percentage rate of patients with complete coverage of all recessions (CRC)

OTHER OUTCOMES:
The depth of gingival sulcus (PD) | 6 months
  Distance from the gingival margin to the deepest point of gingival sulcus

CONTACTS AND LOCATIONS:
Overall Officials: Marta Tanasiewicz, Professor, Study Chair — Department of Conservative Dentistry with Endodontics
Locations (1):
- Department of Periodontal and Oral Mucosa Diseases, Zabrze, Poland